CLINICAL TRIAL: NCT00831688
Title: Phase 3 Study of Efficacy of Local Overpressure Treatment for Meniere's Disease
Brief Title: Efficacy of Local Overpressure Treatment for Meniere's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Responsible Party: Dr. Eike Krause, Klinikum der Universitaet Muenchen, Grosshadern
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Meniere trial 037/05
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Meniere's Disease
Keywords: Meniere; vertigo; overpressure treatment; caloric irrigation; hearing levels; vertigo severity; functional disability scale
MeSH Terms: conditions — Meniere Disease; Vertigo | interventions — Transtympanic Micropressure Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Local overpressure treatment
  Interventions: Device: Meniett(C) device by MedTronic
- 2 (Placebo Comparator): Placebo treatment
  Interventions: Device: placebo treatment

INTERVENTIONS:
Device: Meniett(C) device by MedTronic — pulsed pressure application, up to 12 cm H20 column, 3 times daily for 5 minutes, generated by Meniett device and conducted to middle ear cavity via tympanostomy tube
  Other Names: Meniett
  Arms: 1
Device: placebo treatment — device seemingly identical to active device, manufactured by Medtronic. 3 times daily for 5 minutes.Produces similar sound effect, but without pulsed pressure elevation.
  Other Names: Placebo
  Arms: 2

SUMMARY:
The purpose of this study to date, is that no causal therapy for Meniere's disease has been discovered. Local overpressure treatment for Meniere's disease is a new treatment form that has been shown in animal and human experiments to reduce the endolymphatic hydrops, a condition that is generally believed to be the pathologic hallmark of Meniere's disease. This study analyzes the efficacy of local overpressure treatment by measuring subjective vertigo severity and objective audiovestibular function parameters.

DETAILED DESCRIPTION:
Randomized double-blind controlled trial. Patients with unilateral Meniere's disease that suffer from recurring vertigo attacks are allocated to either a verum or a placebo device and are treated for 4 months. Before during and after the treatment period, subjective and objective audiovestibular function parameters are measured.

ELIGIBILITY:
Inclusion Criteria:

* unilateral definite Meniere's disease according to the AAO-HNS criteria

Exclusion Criteria:

* previous destructive treatment (gentamicin, saccotomy, vestibular neurectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in vertigo score from pre-therapy to post-therapy. (Vertigo score = summation of daily vertigo severity over 4 weeks. Daily vertigo score = a number between = and 4.) | 4 months

SECONDARY OUTCOMES:
Pure tone audiometric thresholds | 4 months
Speech recognition hearing levels | 4 months
Horizontal semicircular canal paresis | 4 Months
Subjective Daily Activity levels (Number between 0 and 4) | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Eike Krause, MD, Principal Investigator — LMU Munich, Department of ENT; Robert Gürkov, MD, Principal Investigator — LMU Munich, Department of ENT
Locations (1):
- Klinik für Hals-Nasen-Ohrenheilkunde, München, Bavaria, Germany